CLINICAL TRIAL: NCT00996983
Title: Phase II Study of Intrathecal Ziconotide for the Treatment of Neuropathic Pain in Patients With Cancer
Brief Title: Safety and Activity Study of Intrathecally Administered Ziconotide for Neuropathic Pain in Patients With Cancer
Acronym: ZIDON
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZIDON; EudraCT number: 2008-005307-26
Record Dates: First submitted 2009-09-30; First posted 2009-10-16 (Estimated); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Pain; Neuropathic Pain; Intractable Pain; Cancer
MeSH Terms: conditions — Pain; Neuralgia; Pain, Intractable; Neoplasms | interventions — ziconotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental)
  Interventions: Drug: ziconotide

INTERVENTIONS:
Drug: ziconotide — intrathecal ziconotide starting at 2.4 micrograms/day, with titration daily to achieve adequate pain control up to maximum dose of 21.6 micrograms/day

SUMMARY:
Neuropathic pain is difficult to control because it is only partially sensitive to opioid analgesics, and requires the addition of other therapies such as antidepressants and epileptics. Ziconotide is a drug that is used to treat neuropathic pain in patients who have had inadequate pain control with prior combination of medicines.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effects and the tolerability of intrathecal ziconotide in cancer patients suffering from severe neuropathic pain not controlled by previous therapies.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of neoplasm
* Neuropathic pain level VASPI > or = 6 (0-10 scale)
* Inadequate pain relief with opioid analgesics and adjuvants
* Age > or = 18 years
* Performance status ECOG 0-2
* Life expectancy at least one month
* Adequate contraception in women of child-bearing potential
* Signed Informed Consent

Exclusion Criteria:

* Use of experimental drugs within previous 30 days
* Pregnancy or lactation
* Contraindication to the use of intrathecal analgesics, including active infection or conditions that could alter the circulation of cerebrospinal fluid
* Presence of cerebral metastasis
* INR > 2
* Contraindication to the use of ziconotide
* Unable or unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2009-09; Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Response rate (> 30% reduction in VASPI) | 48 hours after completion of titration phase

SECONDARY OUTCOMES:
toxicity | daily during drug titration, weekly thereafter
duration of analgesic response | weekly

CONTACTS AND LOCATIONS:
Overall Officials: Arturo Cuomo, M.D., Principal Investigator — NCI Naples, Division of Pain Therapy; Gennaro Russo, M.D., Principal Investigator — NCI Naples, Division of Pain Therapy; Alessandro Morabito, M.D., Principal Investigator — NCI Naples, Clinical Trials Unit
Locations (1):
- Istituto Nazionale dei Tumori , Unita Terapia Antalgica, Napoli, Italy